CLINICAL TRIAL: NCT02850055
Title: Effectiveness Specific Manual Therapy in a Multimodal Physical Therapy Treatment in Patients With Tinnitus and Temporomandibular Joint Disorder.
Brief Title: Effectiveness of Manual Therapy in Patients With Tinnitus and Temporomandibular Joint Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, MARIA JOSE DIAZ ARRIBAS, Tenured University Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MJD_2016
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Tinnitus
Keywords: physiotherapy, Temporomandibular Joint Disorder, tinnitus.
MeSH Terms: conditions — Tinnitus; Temporomandibular Joint Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specific Manual Therapy Group (Experimental): Conventional Physiotherapy and Specific manual therapy, six one hour treatment sessions. An hour for week.
  Interventions: Other: Specific Manual Therapy
- Multimodal Group (Active Comparator): Conventional Physiotherapy, six one hour treatment sessions. An hour for week.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Conventional Physiotherapy — 1. Leaflet care and health habits of the temporomandibular joint.
  2. Program of cranio-cervical and temporomandibular exercises.
  3. Massage of the cervical muscles and self care document for home.
  Other Names: Multimodal Group
  Arms: Multimodal Group
Other: Specific Manual Therapy — 1. Leaflet care and health habits of the temporomandibular joint.
  2. Program of cranio-cervical and temporomandibular exercises.
  3. Massage of the cervical muscles and self care document for home.
  4. Specific manual therapy techniques focusing on the temporomandibular joint and temporomandibular muscles.
  Other Names: Manual Therapy
  Arms: Specific Manual Therapy Group

SUMMARY:
Tinnitus is one of the most prevalent symptoms that causes more disability in patients with temporomandibular disorder (TMD). The present study postulates a possible link between temporomandibular joint (TMJ) and inner ear based on their anatomical, biomechanical and physiological relationship, proposing a physiotherapy treatment for the temporomandibular joint to improve tinnitus. The aim of the study is to evaluate the effectiveness of adding specific manual therapy to a multimodal physiotherapy treatment in patients with tinnitus and temporomandibular disorder.

DETAILED DESCRIPTION:
1. - INTRODUCTION

   Tinnitus is one of the most prevalent symptoms that causes more disability in patients with temporomandibular disorder (TMD).

   According to various studies, the incidence varies between 19-69%, with a 2:1 ratio between women and men, being higher in Western industrialized countries. Frequent conjunction between TMJ problems and tinnitus has led to propose the existence of a link between these two clinical entities. However, the mechanism linking TMD and this otologic symptom is unknown.

   The present study postulates an association based on the anatomical relationship between the TMJ and the inner ear. The ligaments of the inner ear bones are close to TMJ ligaments so the movements of the mandibular condyle may influence on them. The discomallear ligaments (DML) and the anterior mallear ligament (AML) can be considered as intrinsic ligaments of the TMJ.

   TMJ blood supply depends on the tympanic and auricular arteries, and in its innervations are involved nerve branches of the masseter, lateral and temporal/ internal pterygoid, key muscles for the condylar movements (open and close the mouth and lateral movements).

   The hypothesis supporting the link between the TMJ and the tinnitus is that the forced movements of the mandibular condyle produce a ligaments stretching and muscles tension, being the cause of otologic problems such as tinnitus.

   Tinnitus is defined as the perception of a sound that does not exist in the environment. It is often described as "a buzz, a beep, a noise". Most conservative treatments for tinnitus have focused on pharmacological treatments (particularly antidepressants), cognitive-behavioral treatments, medical low strength laser therapies, acupuncture, cranial magnetic stimulation, music therapy and environmental sounds reduction technologies. However, there is controversial evidence on the effectiveness of these techniques given the heterogeneity of protocols and of the response variables.

   Is understood as TMJ pathology, those organic or functional nosological entities affecting the craneomandibular system relationship. They encompass a large number of disorders, not only traumatic, neoplastic, autoimmune or infectious, but also those deriving from dysfunctional alteration of its internal structure, both muscle and joints.

   TMJ disorders with a myofascial or joint dysfunction origin are those whose origin is in myofascial muscle disorders or in joint by mechanical causes. Myofascial trigger points pain, described by Travell and Simons, corresponds to a noninflammatory regional muscle pathology that can occur in any striated muscle of the body. Its main feature is the presence of a hypersensitive area called trigger point, which is present in a palpable taut band of muscle tissue and has the ability to refer pain to distant areas. Joint dysfunction is defined as one in which occurs an abnormal relationship between the joint disk and the condyle, the fossa and the TMJ eminence.

   Many treatments have been applied to the TMJ with varying degrees of evidence: the prevention of bad habits and parafunctions; contract/relax muscles and mental exercises; heat / cold in pain or contracture areas; physiotherapy; psychotherapy; biofeedback techniques with self-relaxation procedures; resting splints, muscle discharge or recapture; transcutaneous electrical nerve stimulation and ultrasound and drug treatment: NSAIDs, analgesics, anxiolytics, hypnotics, muscle relaxants and antidepressants.

   In most cases, the physiotherapy in patients with TMD is focused on myofascial treatment and massage and, at present, in manual therapy (for pain control and improving joint movement). All of this, usually combined with splints or bite plates (for pain control, bruxism and improving occlusion), although there is little evidence supporting their use.

   In relation to myofascial therapy, massage applied on the masticatory muscles, protocols of manual therapy on TMJ, as well as mobilization and manipulation techniques of the upper cervical spine, there is a wide and proven evidence of the improvement occurring in pain, mouth maximum mouth opening and in pressure pain threshold in patients with TMD; although systematic reviews on all manual therapy techniques present a controversial evidence, given the heterogeneity of the studies.

   In the literature review made, it has not been found any paper issuing a proposal or treatment protocol of the TMJ presenting among its main objectives the control of the intensity of TMJ pain and the decrease of disability that tinnitus produces.

   Only one found study proposes a treatment to reduce the intensity of TMJ pain and to improve the disability that tinnitus produces by using a bite splint, without performing a manual intervention therapy and exercises.

   The purpose of the present study is to raise a proposal of treatment with manual therapy and exercise aiming to reduce the disability caused by tinnitus and the intensity of pain and disability caused by the TMD.
2. - JUSTIFICATION

   Tinnitus is one of the most prevalent symptoms that causes more disability in patients with temporomandibular dysfunction (TMD).

   The frequency with which concur the problems of the temporomandibular joint (TMJ) and tinnitus, has led to propose the existence of an association between these two clinical entities.

   The present study postulates the possible link developing an anatomical-pathophysiological hypothesis based on the relationship between TMJ and inner ear, proposing a treatment applied to temporomandibular joint for improving TMJ pain and tinnitus.
3. - HYPOTHESIS AND OBJECTIVES

Hypothesis:

The addition of specific manual therapy techniques (TM) within a multimodal physiotherapy treatment is more effective in improving TMJ pain and disability that causes tinnitus that the isolated application of multimodal treatment.

Objectives:

General:

Evaluate the effectiveness of adding specific manual therapy to a multimodal physical therapy in patients with tinnitus and TMD with a myofascial origin or joint dysfunction.

Specific:

1. Evaluate the effectiveness of adding specific manual therapy to a multimodal physical therapy in patients with tinnitus and TMD in reducing pain intensity and disability caused by TMD.
2. Evaluate the effectiveness of adding specific manual therapy to a multimodal physical therapy in patients with tinnitus and TMD in reducing the intensity of tinnitus and disability caused by tinnitus.
3. Evaluate the effectiveness of adding specific manual therapy to a multimodal physical therapy in patients with tinnitus and TMD in increasing the range of motion of the TMJ.
4. Evaluate the effectiveness of adding specific manual therapy to a multimodal physical therapy in patients with tinnitus and TMD in the painful rise by pressuring the masseter, temporal and lateral pterygoid muscles.
5. Evaluate the effectiveness of adding specific manual therapy to a multimodal physical therapy in patients with tinnitus and TMD in the quality of life, level of anxiety / depression and health.

4. METHODOLOGY

Type of study: randomized and controlled pilot study, multicenter, blinded randomization, patient assessment and data analysis. Treatment characteristics themselves prevent their blinded application.

Location: 3 private consultation rooms of specialized physiotherapy in TMD. Study subjects: 56 patients with temporomandibular dysfunction and tinnitus.

The patient will receive six treatment sessions, two sessions in the first week and a weekly session to complete the intervention. The total duration of the intervention shall be one month. Before starting the study, all patients will be asked to sign an informed consent.

The statistical analysis will be performed using SPSS 22.0 program (IBM statistical software). The average and the standard deviation of quantitative variables will be calculated for the descriptive analysis of the sample if normally distributed.

For the comparative analysis, developed according to the intention to treat:

1. An ANOVA for repeated measure test should be carry out to evaluate the interaction between levels of inter - subject factor (treatment) and the intra- subject (main variables response in time) to be interpreted in case it is significant.
2. To confirm whether this interaction effect is significant, pairwise comparisons will be made of the inter-subjects factor levels (treatment) for each level of main response variables over time using the Bonferroni method.

Limitations of the study - Masking: The nature of the applied treatments prevents masking therapists and patients. This limitation is inherent to the type of treatment evaluated and common with other forms of treatment with similar characteristics, in which therapist should inevitably know the type of treatment that is applied. However, this limitation does not prevent the controlled clinical trials carried out on these technologies from being of higher methodological quality. Thus, in this study, randomization of patients will be blinded, allocation of the random sequence, the assessment of patient evolution and analysis of results.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 65 years old.
* Suffering from tinnitus and temporomandibular dysfunction with a myofascial or joint dysfunction origin: diagnosis of tinnitus attributed to TMD
* In a subacute and chronic phase.

Exclusion Criteria:

* Non signature of the informed consent.
* Patients with a diagnosis of ENT and / or neurological problems from which could arise tinnitus and / or the temporomandibular pain.
* Inability to read, understand and complete questionnaires, read and understand a brochure, or understand and follow verbal commands (e.g. Illiteracy, dementia or blindness).
* Having received physiotherapy in the last 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Intensity of Temporomandibular Joint pain. | At baseline, 1 week post-treatment, and 3 and 6 months post-treatment
  Intensity of TMJ pain (measured by NPRS) at rest.
Change from baseline of tinnitus severity. | At baseline, 1 week post-treatment, and 3 and 6 months post-treatment
  Intensity of tinnitus (measured by VAS) at rest. It will be determined by assessing tinnitus annoyance and tinnitus loudness and the average will be recorded.

SECONDARY OUTCOMES:
Change from baseline degree of tinnitus-related handicap | At baseline, 1 week post-treatment, and 3 and 6 months post-treatment
  Degree of disability caused by tinnitus (measured with the Tinnitus Handicap Inventory (THI).
Change from baseline degree of disability caused by temporomandibular disorder | At baseline, 1 week post-treatment, and 3 and 6 months post-treatment
  Degree of disability caused by temporomandibular disorder (measured by Craniofacial Pain and Disability Inventory (CF-PDI)).
Change from baseline quality of life. | At baseline, 1 week post-treatment, and 3 and 6 months post-treatment
  Quality of life, measured with a previously validated Spanish version of the SF-12 (Short Form Health Survey).
Change from baseline emotional state (depressive symptoms) | At baseline, 1 week post-treatment, and 3 and 6 months post-treatment
  Emotional state of the patient (measured with Beck questionnaire).
Change from baseline pressure pain sensibility | At baseline, 1 week post-treatment, and 3 and 6 months post-treatment
  Pain sensibility to pressure (measured with an algometer) in the masseter, temporal and lateral pterygoid muscles (over the TMJ).
Change from baseline range of motion | At baseline, 1 week post-treatment, and 3 and 6 months post-treatment
  Range of motion of the temporomandibular joint in the mouth opening and bilateral excursion movements (measured in millimetres)

CONTACTS AND LOCATIONS:
Overall Officials: María J Díaz, Professor, Study Director — Physiotherapy Professor
Locations (1):
- María José Díaz Arribas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calixtre LB, Moreira RF, Franchini GH, Alburquerque-Sendin F, Oliveira AB. Manual therapy for the management of pain and limited range of motion in subjects with signs and symptoms of temporomandibular disorder: a systematic review of randomised controlled trials. J Oral Rehabil. 2015 Nov;42(11):847-61. doi: 10.1111/joor.12321. Epub 2015 Jun 7. PMID 26059857
- [Background] Langguth B. Treatment of tinnitus. Curr Opin Otolaryngol Head Neck Surg. 2015 Oct;23(5):361-8. doi: 10.1097/MOO.0000000000000185. PMID 26261868
- [Background] Plein CT, Harounian J, Floyd E, Irizarry R, Ferzli G, Kidwai S, Rosenfeld RM. A Systematic Review of Eligibility and Outcomes in Tinnitus Trials: Reassessment of Tinnitus Guideline. Otolaryngol Head Neck Surg. 2016 Jan;154(1):24-32. doi: 10.1177/0194599815608160. Epub 2015 Oct 12. PMID 26459245
- [Background] Sencimen M, Yalcin B, Dogan N, Varol A, Okcu KM, Ozan H, Aydintug YS. Anatomical and functional aspects of ligaments between the malleus and the temporomandibular joint. Int J Oral Maxillofac Surg. 2008 Oct;37(10):943-7. doi: 10.1016/j.ijom.2008.07.003. Epub 2008 Sep 2. PMID 18768297
- [Background] Al-Ani MZ, Davies SJ, Gray RJ, Sloan P, Glenny AM. WITHDRAWN: Stabilisation splint therapy for temporomandibular pain dysfunction syndrome. Cochrane Database Syst Rev. 2016 Jan 4;2016(1):CD002778. doi: 10.1002/14651858.CD002778.pub3. PMID 26727210
- [Background] Ebrahim S, Montoya L, Busse JW, Carrasco-Labra A, Guyatt GH; Medically Unexplained Syndromes Research Group. The effectiveness of splint therapy in patients with temporomandibular disorders: a systematic review and meta-analysis. J Am Dent Assoc. 2012 Aug;143(8):847-57. doi: 10.14219/jada.archive.2012.0289. PMID 22855899
- [Background] La Touche R, Fernandez-de-las-Penas C, Fernandez-Carnero J, Escalante K, Angulo-Diaz-Parreno S, Paris-Alemany A, Cleland JA. The effects of manual therapy and exercise directed at the cervical spine on pain and pressure pain sensitivity in patients with myofascial temporomandibular disorders. J Oral Rehabil. 2009 Sep;36(9):644-52. doi: 10.1111/j.1365-2842.2009.01980.x. Epub 2009 Jul 14. PMID 19627454
- [Background] La Touche R, Paris-Alemany A, Mannheimer JS, Angulo-Diaz-Parreno S, Bishop MD, Lopez-Valverde-Centeno A, von Piekartz H, Fernandez-Carnero J. Does mobilization of the upper cervical spine affect pain sensitivity and autonomic nervous system function in patients with cervico-craniofacial pain?: A randomized-controlled trial. Clin J Pain. 2013 Mar;29(3):205-15. doi: 10.1097/AJP.0b013e318250f3cd. PMID 22874091
- [Background] Armijo-Olivo S, Pitance L, Singh V, Neto F, Thie N, Michelotti A. Effectiveness of Manual Therapy and Therapeutic Exercise for Temporomandibular Disorders: Systematic Review and Meta-Analysis. Phys Ther. 2016 Jan;96(1):9-25. doi: 10.2522/ptj.20140548. Epub 2015 Aug 20. PMID 26294683
- [Background] Attanasio G, Leonardi A, Arangio P, Minni A, Covelli E, Pucci R, Russo FY, De Seta E, Di Paolo C, Cascone P. Tinnitus in patients with temporo-mandibular joint disorder: Proposal for a new treatment protocol. J Craniomaxillofac Surg. 2015 Jun;43(5):724-7. doi: 10.1016/j.jcms.2015.02.009. Epub 2015 Mar 12. PMID 25868942
- [Background] La Touche R, Pardo-Montero J, Gil-Martinez A, Paris-Alemany A, Angulo-Diaz-Parreno S, Suarez-Falcon JC, Lara-Lara M, Fernandez-Carnero J. Craniofacial pain and disability inventory (CF-PDI): development and psychometric validation of a new questionnaire. Pain Physician. 2014 Jan-Feb;17(1):95-108. PMID 24452650
- [Background] Vilagut G, Valderas JM, Ferrer M, Garin O, Lopez-Garcia E, Alonso J. [Interpretation of SF-36 and SF-12 questionnaires in Spain: physical and mental components]. Med Clin (Barc). 2008 May 24;130(19):726-35. doi: 10.1157/13121076. Spanish. PMID 18570798
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomized trials. Ann Intern Med. 2010 Jun 1;152(11):726-32. doi: 10.7326/0003-4819-152-11-201006010-00232. Epub 2010 Mar 24. PMID 20335313
- [Background] Knol MJ, Groenwold RH, Grobbee DE. P-values in baseline tables of randomised controlled trials are inappropriate but still common in high impact journals. Eur J Prev Cardiol. 2012 Apr;19(2):231-2. doi: 10.1177/1741826711421688. No abstract available. PMID 22512015
- [Background] Kalamir A, Bonello R, Graham P, Vitiello AL, Pollard H. Intraoral myofascial therapy for chronic myogenous temporomandibular disorder: a randomized controlled trial. J Manipulative Physiol Ther. 2012 Jan;35(1):26-37. doi: 10.1016/j.jmpt.2011.09.004. Epub 2011 Nov 10. PMID 22079052
- [Background] Gomes CA, Politti F, Andrade DV, de Sousa DF, Herpich CM, Dibai-Filho AV, Gonzalez Tde O, Biasotto-Gonzalez DA. Effects of massage therapy and occlusal splint therapy on mandibular range of motion in individuals with temporomandibular disorder: a randomized clinical trial. J Manipulative Physiol Ther. 2014 Mar-Apr;37(3):164-9. doi: 10.1016/j.jmpt.2013.12.007. Epub 2014 Jan 3. PMID 24387891
- [Derived] Delgado de la Serna P, Plaza-Manzano G, Cleland J, Fernandez-de-Las-Penas C, Martin-Casas P, Diaz-Arribas MJ. Effects of Cervico-Mandibular Manual Therapy in Patients with Temporomandibular Pain Disorders and Associated Somatic Tinnitus: A Randomized Clinical Trial. Pain Med. 2020 Mar 1;21(3):613-624. doi: 10.1093/pm/pnz278. PMID 31665507